CLINICAL TRIAL: NCT04192058
Title: Effect of Transcranial Direct-current Stimulation in Homeostastic and Hedonistic Mechanisms of Eating Behavior in Women With Fibromyalgia
Brief Title: Effect of Transcranial Direct-current Stimulation in Eating Behavior of Women With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-0237
Record Dates: First submitted 2019-10-31; First posted 2019-12-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia; Food Addiction
Keywords: polymorphism Taq1A; tDCS; dopamine; eating behavior
MeSH Terms: conditions — Fibromyalgia; Food Addiction; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham tDCS (Sham Comparator): For sham treatment we will use the same assembly as the active ETCC. However, we will apply the current for 30s at the start of the stimulation session and 30s at the end of the session.
  Interventions: Device: Sham transcranial direct current stimulation (tDCS)
- active tDCS (Experimental): The anode will be positioned over the left hemisphere at C3 while the cathode will be positioned over the contralateral hemisphere F3. During active stimulation a 2.0mA current released by a 35 cm2 electrode will be used for 20 min. The position of the electrodes will be performed based on a 10-20 system according to the international EEG unit system, with the location of the electrodes at C3 and F3, respectively.
  Interventions: Device: Active transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Sham transcranial direct current stimulation (tDCS) — For sham treatment we will use the same assembly as the active ETCC. However, we will apply the current for 30s at the start of the stimulation session and 30s at the end of the session.
  Arms: sham tDCS
Device: Active transcranial direct current stimulation (tDCS) — Transcranial direct current stimulation (tDCS) it is a therapeutic method that modulates membrane potential, where anodic stimuli induce cortical excitability and cathodic stimuli reduce it. The position of the electrodes will be performed based on a 10-20 system according to the international EEG unit system, with the location of the electrodes at C3 and F3, respectively. The anode will be positioned over the left hemisphere at C3 while the cathode will be positioned over the contralateral hemisphere F3. During active stimulation a 2.0mA current released by a 35 cm2 electrode will be used for 20 min.
  Arms: active tDCS

SUMMARY:
Introduction: Fibromyalgia (FM) is a syndrome characterized by generalized musculoskeletal pain, fatigue, non-repairing sleep, cognitive changes, depressive symptoms and other correlates of autonomic dysfunction. A high prevalence of overweight in patients with fibromyalgia is observed, about 80% according to current data, which affects the course and prognosis of the disease, besides overburdening health costs and further compromising quality of life. life of these patients. Evidence shows possible pathophysiological pathways shared by these two pathologies, as well as aspects related to food behavior. It is known that dopaminergic neurotransmission is altered in both, suggesting an increase in the sensitivity or density of D2 dopamine receptors. Non-pharmacological options for pain management and dysfunctional eating behavior include the important contribution of neuromodulatory techniques of non-invasive cerebral stimulation, such as transcranial direct current stimulation (tDCS), which aims to increase resisting hyperpalatable foods and reducing caloric intake. Objectives: To evaluate the association between dopamine receptor-2 (DRD2) Taq1A allele A1 polymorphism (rs1800497) and to observe the possible effect of tDCS on the dorsolateral prefrontal cortex (DLPFC) on homeostatic and hedonistic aspects of eating behavior in women with FM. Methods: A randomized, double blind, parallel group, controlled trial with simulated treatment will be performed. Will be included in the study women literate, right-handed, with confirmed diagnosis of FM. The evaluation will be done through questionnaires on pain and eating behavior, anthropometric evaluation and biochemical measurements. The intervention will take place through active or simulated home for 4 weeks. Perspectives: To evaluate dysfunctional neuroplastic changes in eating behavior and biological markers and also to serve as a basis for future effective treatment strategies through neuromodulation and nutritional counseling.

DETAILED DESCRIPTION:
A randomized, double-blind, parallel-group controlled trial with sham treatment will be conducted in fibromyalgia patients to assess aspects of eating behavior.

ELIGIBILITY:
Inclusion criteria:

* Right-handers who can read and write,
* Confirmed diagnosis of FM
* Pain score of six or more on the Numerical Pain Scale (SPN 0-10) on most days of the last 3 months.

Exclusion criteria:

Living outside the Greater Porto Alegre area and pregnancy. Contraindications to EMT and ETCC: metallic implant in the brain; medical devices implanted in the brain, cardiac pacemaker; cochlear implant; history of alcohol or drug abuse in the last 6 months; neurological disorders; hx of head trauma or neurosurgery; decompensated systemic diseases, and chronic inflammatory diseases (lupus, rheumatoid arthritis, Sjogren's syndrome, Reiter's syndrome); uncompensated hypothyroidism; personal history of cancer, past or under treatment. Weight loss use and bariatric surgery.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-11-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Three Factor Eating Questionnaire 21 | 6 mouths
  TFE-Q was developed by Stunkard and Messic (1985) to access three dimensions of human eating behavior: Cognitive Restriction (CR), Eating Disorder (AD) and Emotional Eating (AE). Originally made up of 51 items and reduced in the TFEQ-18, TFEQ-18, TFEQ-21 versions. We will use the TFEQ-21. The average obtained from the sum of the questions for each domain was converted to a scale ranging from 0 to 100.
  Evaluates dysfunctional eating behavior. Cognitive restriction: limitation of food intake for weight control; Uncontrolled Food: Tendency to lose control over eating from hunger or when exposed to external environments, even in the absence of physiological hunger; Emotional Eating: Susceptible to eating in response to emotional stress or negative mood.

SECONDARY OUTCOMES:
weight | up to 2 weeks
  measured by scale
waist circumference. | up to 2 weeks
  measured by measuring tape
State and Trait Food-Cravings Questionnaires (FCQ-s e FCQ-t) | 6 mouths
  - FCQ-T consists of 39 statements and was developed to access food cravings aspects over time and in various situations, considering them as a (usual) trait behavior of the respondent.
  Higher scores in this questionnaire are related to a more exaggerated eating.
  - FCQ-S is composed of 15 statements and is a tool sensitive to changes in contextual, psychological and physiological states in response to specific situations (such as stressful events or food deprivation), considering the food craving as a (sporadic) state behavior of the respondent.
  Higher scores in this questionnaire are associated with greater food deprivation, negative eating-related experiences and a greater susceptibility to triggers that lead to eating.
  Totals of both tools for the full subscales and their dimensions are calculated by adding the corresponding scores of each statement.
Hunger and satiety diary | up to 24 hours
  Hunger and satiety measured by the 100 mm Analog-Visual Scale (VAS), whose zero corresponds to the absence of hunger or appetite and 100 mm hunger or maximum appetite. Patients should report hunger, hunger or satiety for most of the last 24 hours.
Appetite Diary | up to 24 hours
  Appetite measured by means of the 100 mm Analog-Visual Scale (VAS), whose zero corresponds to the absence of appetite and 100 mm or maximum appetite. Patients should report nonspecific appetite for sweet or salty most of the last 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, Md PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Wolnei Caumo, Porto Alegre

IPD SHARING:
Plan to Share IPD: No